CLINICAL TRIAL: NCT01519414
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Study of ARQ 197 (Tivantinib) in Men With Asymptomatic or Minimally Symptomatic Metastatic Castrate Resistant Prostate Cancer
Brief Title: Tivantinib in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-00237; NCI-2012-00237 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000721410; OSU11132; OSU-11132; OSU 11132 (Other: Ohio State University Comprehensive Cancer Center); 8986 (Other: CTEP); N01CM00070 (NIH); N01CM00071 (NIH); N01CM00100 (NIH); N01CM62207 (NIH); P30CA016058 (NIH); U01CA062491 (NIH)
Record Dates: First submitted 2012-01-25; First posted 2012-01-27 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Hormone-Resistant Prostate Cancer; Prostate Adenocarcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ARQ 197

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (tivantinib) (Experimental): Patients receive tivantinib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Tivantinib
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may crossover to Arm I.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Optional correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Drug: Tivantinib — Given PO
  Other Names: ARQ 197; ARQ-197; c-Met Inhibitor ARQ 197
  Arms: Arm I (tivantinib)

SUMMARY:
This randomized phase II trial studies how well tivantinib works compared to placebo in treating patients with metastatic prostate cancer. Tivantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine progression-free survival (PFS) in men with minimally symptomatic or asymptomatic metastatic, castrate-resistant, chemotherapy-naïve prostate cancer treated with ARQ 197 (tivantinib).

SECONDARY OBJECTIVES:

I. To determine the prostate-specific antigen (PSA) response rate at 12 weeks in men with metastatic, castrate-resistant, chemotherapy-naïve prostate cancer treated with ARQ 197.

II. To determine the radiographic response rate at 12 weeks based on Response Evaluation Criteria in Solid Tumors (RECIST) criteria on computed tomography (CT) scans and stability of bone lesions on bone scan in castrate-resistant, chemotherapy-naïve prostate cancer treated with ARQ 197.

III. To determine the proportion of patients who are progression-free at 12 weeks.

IV. To assess safety and tolerability in patients treated with ARQ 197 using the National Institute of Cancer (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 grading of toxicities.

TERTIARY OBJECTIVES:

I. Evaluate markers of bone turnover. (Exploratory)

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive tivantinib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Arm II: Patients receive placebo PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may crossover to Arm I.

After completion of study treatment, patients are followed up every 3 months for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented adenocarcinoma of the prostate with progressive systemic disease (either rising PSA or progression of disease on CT scan or magnetic resonance imaging [MRI] or bone scan) despite castrate levels of testosterone due to orchiectomy or luteinizing hormone-releasing hormone (LHRH) agonist or antagonist; castrate levels of testosterone must be maintained throughout the study
* Evidence of metastatic disease on CT or bone imaging
* Patients must have demonstrated evidence of progressive disease since the most recent change in therapy; progressive disease is defined as any one of the following (measurable disease, bone scan, or PSA progression):

  * Measurable disease progression: objective evidence of increase > 20% in the sum of the longest diameters (LD) of target lesions from the time of maximal regression or the appearance of one or more new lesions
  * Bone scan progression: appearance of two or more new lesions on bone scan attributable to prostate cancer will constitute progression
  * PSA progression: two successive rises from baseline PSA separated at least by one week with the last value >= 2 ng/mL
* Asymptomatic or minimally symptomatic from prostate cancer - no symptoms attributed to prostate cancer greater than grade I using NCI CTCAE version 4.0 grading of toxicities
* Secondary hormonal therapies (e.g., abiraterone acetate, flutamide, estrogen) must be discontinued for at least 4 weeks prior to study enrollment unless the duration of the therapy was less than 8 weeks and there was no demonstrated decrease in PSA
* Secondary hormonal therapies with bicalutamide or nilutamide must be discontinued for 6 weeks unless duration of therapy was less than 8 weeks and there was no demonstrated PSA decrease
* Prior abiraterone (or investigational anti-androgen) use is allowed; these too will need to be discontinued at least 4 weeks prior to study enrollment
* PSA prior to treatment must be >= 2 ng/ml
* Castrate testosterone level (< 50 ng/dL)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* No prior chemotherapy unless utilized in neoadjuvant/adjuvant setting and must have completed > 6 months prior to enrollment
* Four weeks since major surgery or radiation therapy
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.0 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 40 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must have signed an informed consent document stating that they understand the investigational nature of the proposed treatment
* Men and any female partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation and for additional 2 months after finishing therapy; should a patient's sexual partner become pregnant or suspect she is pregnant while patient is participating in this study, he should inform the treating physician immediately
* Bisphosphonate or denosumab therapy is permitted provided patients began therapy prior to registration and that they continue them as per the manufacturer's guidelines and/or per institutional practice; patients not taking ongoing bisphosphonate or denosumab therapy will not be permitted to start such therapy until they have completed 12 weeks of study treatment
* Patients must be able to swallow pills to participate in the study

Exclusion Criteria:

* Patients who have radiotherapy within 4 weeks or chemotherapy prior to entering the study or those who have not recovered (resolution to grade 1) from adverse events due to agents administered more than 4 weeks earlier; neoadjuvant/adjuvant chemotherapy for local disease is allowed if greater than 6 months have elapsed
* Previous hepatocyte growth factor receptor (C-MET) inhibitor treatment (either monoclonal antibody to C-MET or human growth factor [HGF] or small molecule inhibitory to C-MET)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition ARQ 197
* Caution should be used with patients receiving inhibitors of cytochrome P450 family 2, subfamily C, polypeptide 19 (CYP2C19) and strong inhibitors of cytochrome P450 family 3, subfamily A, polypeptide4 (CYP3A4); additional hematologic testing will be advised if the medication cannot be substituted
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or known psychiatric illness/social situations that would limit compliance with study requirements
* Known brain metastasis
* Current, recent (within 4 weeks of the first study drug administration), or concurrent planned participation in another investigational therapeutic study
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers are not to be registered; patients are not considered to have a "currently active" malignancy if they have completed therapy and are now considered to be at less than 30% risk for relapse (by their physician)
* Patients may continue on a daily multi-vitamin and calcium/vitamin D supplements; all other herbal, alternative, and food supplements (i.e., PC-SPES, Saw Palmetto, St. John wort, etc.) must be discontinued before registration
* New York Heart Association (NYHA) class III or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to initial treatment
* History of severely impaired lung function
* Baseline electrocardiogram (ECG) abnormalities including first degree (PR interval > 210 ms), second degree, or third degree heart block (exception: patients with pacemakers may be enrolled); QRS prolongation or bundle branch block (QRS >= 120 ms), or QT prolongation (per institutional standard of care: Fridericia corrected QT interval [QTcF] or Bazett corrected QT interval [QTcB] >= 470 ms); other ECG abnormalities will need consideration by the treating investigator and enrollment is up to his/her discretion
* Presence of non-healing wound, active ulcer, or untreated bone fracture
* Known diabetics that have poorly controlled diabetes mellitus (glycated hemoglobin [HbA1c] >= 8.0%) or fasting glucose level >= 189 mg/dL (diabetic patient); patients may be potentially eligible once anti-diabetic agent(s) are either added or titrated to control their diabetes mellitus
* Active liver disease (AST or ALT >= 2.0 times the upper limit of normal [ULN] or total bilirubin >= institutional ULN) or gallbladder disease; patients with known liver cirrhosis or severe hepatic impairment (Child-Pugh Class C) will also be excluded
* A known history of human immunodeficiency virus (HIV) seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of ARQ 197 (e.g., uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or significant small bowel resection)
* Patients with an active bleeding diathesis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-01-11 (Actual); Primary Completion 2015-08-18 (Actual); Study Completion 2015-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Monk, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (20):
- United States (20):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Michael Reese Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc - Jefferson Boulevard, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - University of Maryland Saint Joseph Medical Center, Towson, Maryland
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Tivantinib): Patients receive tivantinib 360 mg (3 * 120 mg tablets) po BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm II (Placebo): Patients receive matched placebo (3 tablets) po BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may crossover to Arm I.
- Crossover From Placebo to Tivantinib: Patients who were originally assigned to placebo and experience disease progression will be allowed to crossover and take ARQ 197. The treatment plan, duration of therapy, criteria for progression and follow-up will be the same as described above for men originally assigned to ARQ 197.
Period: Pre Cross-over
Arm/Group | Arm I (Tivantinib) | Arm II (Placebo) | Crossover From Placebo to Tivantinib
Started | 52 | 26 | 0
Completed | 52 | 26 | 0
Not Completed | 0 | 0 | 0
Period: Post Cross-over
Arm/Group | Arm I (Tivantinib) | Arm II (Placebo) | Crossover From Placebo to Tivantinib
Started | 52 | 14 | 12
Completed | 52 | 14 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Tivantinib) | Arm II (Placebo) | Total
Number analyzed (Participants) | 52 | 26 | 78
Age, Continuous [Median (Full Range); unit: years] | 67 [43 to 84] | 66.5 [48 to 85] | 67 [43 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 52 | 26 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 49 | 20 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: patients]
  United States | 52 | 26 | 78

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Based on the RECIST Criteria
Description: The progression-free survival distributions between the two arms will be compared using log-rank tests. Progression-free survival curves will be constructed using the Kaplan-Meier product limit method, and additional analyses will be done using the Cox proportional hazards model.
Time Frame: Time from study entry to the date of documented progression and/or death, assessed up to 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Tivantinib) | Arm II (Placebo)
Number analyzed (Participants) | 52 | 26
months | 5.5 [3.2 to 8.0] | 3.7 [2.7 to 5.4]
Statistical Analysis 1: Comparison: Arm I (Tivantinib) vs Arm II (Placebo); Test type: Other; p = 0.02, Log Rank

2. Secondary Outcome: Changes in PSA Levels
Description: Evaluated and patterns graphically explored through waterfall plots.
Time Frame: Baseline to 12 weeks
Measure: Median (Full Range); unit: percentage change from baseline
Arm/Group | Arm I (Tivantinib) | Arm II (Placebo)
Number analyzed (Participants) | 52 | 26
percentage change from baseline | 140.1 [-9.0 to 5768.1] | 301.5 [-3.3 to 3254.4]

3. Secondary Outcome: Proportion of Patients Who Respond
Description: An assumed binomial distribution used. Summarized with their corresponding 95% binomial confidence intervals and compared in an exploratory manner between the two treatment arms. Dichotomized outcomes of response will be descriptively summarized and graphically evaluated using bar graphs.
Time Frame: At 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Arm I (Tivantinib): Arm I: Patients receive tivantinib 360 mg (3 * 120 mg tablets) po BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm II (Placebo): Patients receive placebo PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may crossover to
Arm/Group | Arm I (Tivantinib) | Arm II (Placebo) | Crossover From Placebo to Tivantinib
Number analyzed (Participants) | 52 | 26 | 12
percentage of patients | 1.9 [0.05 to 10.26] | 0 [0 to 0] | 8.3 [0.2 to 38.5]

4. Secondary Outcome: PSA Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: up to 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm I (Tivantinib) | Arm II (Placebo) | Crossover From Placebo to Tivantinib
Number analyzed (Participants) | 52 | 26 | 12
percentage of patients | 1.9 [0.05 to 10.26] | 0 [0 to 0] | 8.3 [0.2 to 38.5]

5. Secondary Outcome: Incidence of Adverse Events Graded as 3, 4, or 5 Per NCI CTCAE Version 4.0
Description: Fisher's exact tests will be used to quantitatively compare the incidence of severe as well as specific toxicities of interest between the treatment arms and graphically assessed differences in maximum grades observed for toxicities between the arms.
Time Frame: Up to 1 year
Population: Adverse events graded as 3, 4 or 5 per NCI CTCAE version 4 (regardless of attribution)
Measure: Number; unit: patients
Arm/Group | Arm I (Tivantinib) | Arm II (Placebo) | Crossover From Placebo to Tivantinib
Number analyzed (Participants) | 52 | 26 | 12
patients
  Acute coronary syndrome | 1 | 0 | 0
  Alkaline phosphatase increased | 0 | 0 | 2
  Anemia | 3 | 0 | 2
  Back pain | 1 | 1 | 1
  Confusion | 0 | 2 | 0
  Cataract | 1 | 0 | 0
  Death NOS | 1 | 0 | 1
  Dehydration | 0 | 2 | 1
  Dizziness | 0 | 1 | 0
  Duodenal ulcer | 1 | 0 | 0
  Dyspnea | 0 | 1 | 0
  Enterocolitis infectious | 0 | 1 | 0
  Fall | 0 | 1 | 0
  Fatigue | 2 | 0 | 0
  Febrile neutropenia | 1 | 0 | 0
  Gait disturbance | 0 | 1 | 0
  Generalized muscle weakness | 0 | 1 | 0
  Hypertension | 1 | 0 | 0
  Hypokalemia | 0 | 1 | 0
  Hyponatremia | 1 | 0 | 0
  Hypotension | 0 | 1 | 0
  Hypoxia | 1 | 1 | 0
  Infections and infestations - Other, specify | 1 | 0 | 0
  Lymph gland infection | 1 | 0 | 0
  Lymphocyte count decreased | 2 | 2 | 2
  Musculoskeletal and connective tissue disorder - O | 0 | 1 | 0
  Neoplasms benign, malignant and unspecified (incl | 1 | 1 | 0
  Nervous system disorders - Other, specify | 0 | 1 | 0
  Neutrophil count decreased | 2 | 0 | 2
  Platelet count decreased | 1 | 0 | 0
  Pleural effusion | 0 | 0 | 1
  Productive cough | 0 | 0 | 1
  Sinus bradycardia | 3 | 0 | 0
  Sinus tachycardia | 0 | 1 | 0
  Syncope | 0 | 2 | 0
  Thromboembolic event | 0 | 1 | 0
  Tumor pain | 1 | 0 | 0
  Upper respiratory infection | 0 | 1 | 0
  Urinary tract obstruction | 0 | 0 | 1
  White blood cell decreased | 2 | 0 | 2

6. Other Pre Specified Outcome: Radiographic Response Rate Based on RECIST Criteria
Description: Summarized with their corresponding 95% binomial confidence intervals and compared in an exploratory manner between the two treatment arms. Dichotomized outcomes of response will be descriptively summarized and graphically evaluated using bar graphs.
Time Frame: Up to 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Arm II (Placebo): Arm II: Patients receive matched placebo (3 tablets) po BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may crossover to Arm I.
Arm/Group | Arm I (Tivantinib) | Arm II (Placebo) | Crossover From Placebo to Tivantinib
Number analyzed (Participants) | 52 | 26 | 12
percentage of patients | 1.9 [0.05 to 10.26] | 0 [0 to 0] | 8.3 [0.2 to 38.5]

7. Other Pre Specified Outcome: Change in Bone Specific Alkaline Phosphatase (BSAP) in Serum
Description: BSAP will first be descriptively summarized by treatment group and also evaluated using graphical analyses to assess potential patterns over time and see if changes in bone resorption differ between those who are progression-free at 12 weeks vs. not after treatment with tivantinib. The potential impact of early changes in these markers on PFS using Cox regression models will be also explored.
Time Frame: Baseline to up to 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Markers of Bone Turnover in Urine
Description: NTx and CTX will first be descriptively summarized by treatment group and also evaluated using graphical analyses to assess potential patterns over time and see if changes in bone resorption differ between those who are progression-free at 12 weeks vs. not after treatment with tivantinib. The potential impact of early changes in these markers on PFS using Cox regression models will be also explored.
Time Frame: Baseline to up to 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: The National Cancer Institutes (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting.
Arm/Group | Arm I (Tivantinib) | Arm II (Placebo) | Crossover From Placebo to Tivantinib
All-Cause Mortality (participants affected / at risk) | 7/52 | 4/26 | 0/12
Serious Adverse Events (participants affected / at risk) | 19/52 | 22/26 | 5/12
Other Adverse Events (participants affected / at risk) | 52/52 | 26/26 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Tivantinib) (N=52) | Arm II (Placebo) (N=26) | Crossover From Placebo to Tivantinib (N=12)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Tivantinib) (N=52) | Arm II (Placebo) (N=26) | Crossover From Placebo to Tivantinib (N=12)
Anemia (Blood and lymphatic system disorders) | 23 (23) | 12 (12) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 11 (11) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 2 (2) | 3 (3) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Flashing lights (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 14 (14) | 7 (7) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 4 (4) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (9) | 5 (5) | 3 (3)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 2 (2)
Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 5 (5) | 2 (2) | 1 (1)
Edema trunk (General disorders) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 30 (30) | 11 (11) | 7 (7)
Fever (General disorders) | 1 (1) | 1 (1) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 2 (2) | 2 (2) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0)
Neck edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 5 (5) | 7 (7) | 2 (2)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (7) | 2 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 8 (8) | 5 (5) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 13 (13) | 3 (3) | 2 (2)
Creatinine increased (Investigations) | 7 (7) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 11 (11) | 6 (6) | 4 (4)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (5) | 0 (0) | 5 (5)
Platelet count decreased (Investigations) | 3 (3) | 2 (2) | 1 (1)
Weight gain (Investigations) | 2 (2) | 0 (0) | 0 (0)
Weight loss (Investigations) | 4 (4) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 12 (12) | 1 (1) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 17 (17) | 5 (5) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (9) | 3 (3) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 11 (11) | 3 (3) | 3 (3)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 13 (13) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (13) | 11 (11) | 2 (2)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 5 (5) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 4 (4) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 4 (4) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Hot flashes (Vascular disorders) | 5 (5) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less